CLINICAL TRIAL: NCT03555279
Title: PHAT Life: Peer Versus Adult-Led HIV Prevention for Juvenile Offenders
Acronym: PHATLife
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Geri Donenberg, Professor, Departments of Medicine and Psychology, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-0936; 1R01MD010433 (NIH)
Record Dates: First submitted 2018-05-18; First posted 2018-06-13 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: HIV/AIDS
Keywords: HIV Prevention; Juvenile Justice; Sexual Health; Evidence Based Intervention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probation Staff (PS) Facilitator (Experimental): The PHAT Life: Preventing HIV/AIDS Among Teens--PS Arm intervention is delivered by Probation Staff working at the intervention site. Dosage is 8 2-hour sessions delivered over two weeks.
  Interventions: Behavioral: PHAT Life: Preventing HIV/AIDS Among Teens--PS Arm
- Youth Representative (YR) Facilitator (Experimental): The PHAT Life: Preventing HIV/AIDS Among Teens--YR Arm intervention is delivered by young adults who were formally in the juvenile justice system. Dosage is 8 2-hour sessions delivered over two weeks.
  Interventions: Behavioral: PHAT Life: Preventing HIV/AIDS Among Teens--YR Arm

INTERVENTIONS:
Behavioral: PHAT Life: Preventing HIV/AIDS Among Teens--PS Arm — HIV Prevention Behavioral Health Intervention delivered by Probation Staff
  Arms: Probation Staff (PS) Facilitator
Behavioral: PHAT Life: Preventing HIV/AIDS Among Teens--YR Arm — HIV Prevention Behavioral Health Intervention delivered by Youth Representatives
  Arms: Youth Representative (YR) Facilitator

SUMMARY:
This application proposes a 2-arm randomized controlled trial comparing the impact of PHAT Life on 350 13-17 year-old offenders' risky sex, STI, substance use, and theoretical mediators when delivered by Youth Representatives (YR) vs. probation staff (PS). 100 facilitators will be recruited to deliver the intervention and participate in the research.

DETAILED DESCRIPTION:
The main objectives of the proposed study are to compare the effectiveness, cost-effectiveness, and sustainability of Youth Representative-led vs. probation staff-led PHAT Life in a real-world juvenile probation setting. The Specific Aims of this study are:

1. To conduct a methodologically-rigorous 2-arm trial comparing the impact of PHAT Life on 350 13-17 year-old offenders' risky sex, STI, substance use, and theoretical mediators when delivered by Youth Representatives (YR) vs. probation staff (PS).
2. To compare the costs and cost-effectiveness of 100 YR-led vs. PS-led PHAT Life with respect to the acquisition of incident STI.

We hypothesize: (a) Compared to teens in PS-led groups, we expect teens in YR-led groups to report less risky sex and substance use at 6-month follow-up, to demonstrate greater improvement on theoretical mediators of risk, and to have fewer incident STI infections; (b) We expect YR-led PHAT Life to cost less and be more cost-effective than PS-led PHAT Life.

ELIGIBILITY:
Inclusion Criteria:

a) male or female gender; b) remanded to a probation program; c) 13-17 years old; d) adolescent is fluent in English; e) are not wards of the Department of Child and Family Services (DCFS); and f) they have not already received the PHAT Life intervention.

Exclusion Criteria:

a) are unable to understand the consent/assent process; b) do not speak English, because instruments are normed for English speakers; c) do not assent; d) legal guardians do not consent to teens' participation; e) are not 13 -17 years old; f) are not on probation or remanded to a probation program; g) are wards of the Department of Child and Family Services (DCFS); and h) they have already received the PHAT Life intervention.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 218 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Change in HIV/STI Risk Behaviors at 6 months | Baseline and 6-months
  AIDS Risk Behavior Assessment (ARBA) A computer-assisted structured interview of self-reported sexual behavior and drug use derived from five well-established measures. The outcomes include ever had sex, condom use, number of partners, sex while using drugs and/or alcohol.

SECONDARY OUTCOMES:
Change in HIV/AIDS/STI Knowledge, Attitudes, Beliefs, and Behavioral Skills at 6 | Baseline and 6-months
  Survey measuring knowledge regarding transmission routes, misconceptions about transmission, and risk-reduction strategies; attitudes and beliefs including peer norms, intentions to prevent HIV/AIDS/STI, attitudes towards preventive actions, and beliefs about condom use; as well as self-efficacy to prevent transmission, apply condoms, and negotiate with a partner.
Change in mental health symptoms at 6 months | Baseline and 6-months
  The Youth Self Report (YSR) is a widely-used and validated measure of child behavior problems that generates raw and T-scores for internalizing and externalizing syndromes as well as narrow-band problems (e.g., delinquency, anxiety, depression).
Change in Partner Sexual Communication at 6 months | Baseline and 6-months
  Questionnaire in which participants indicate whether they ever talked to their romantic or dating partners and sexual partners about a list of sexual topics, how often they discussed them, and whether they talk was open and comfortable. Items were adapted from the Sexual Risk Behavior Questionnaire.
Change in Relationship dynamics at 6 months | Baseline and 6-months
  The Sexual Relationship Power Scale (SRPS) measures perceptions of relationship control and decision-making dominance. It has good internal consistency and predictive and constructed validity.
Change in trauma symptoms and violence exposure at 6 months | Baseline and 6-months
  The UCLA PTSD Index will measure exposure to trauma and violence.
Change in peer influences at 6 months | Baseline and 6-months
  The Peer Convention Behavior Questionnaire will measure peer support of risky behavior, peer norms, and peer pressure and teens' association with prosocial peers.
Change in parental Influences at 6 months | Baseline and 6-months
  The Parenting Style Questionnaire (PSQ) measures parental supervision, monitoring, and permissiveness.
Change in parental communication at 6 months | Baseline and 6-months
  The Parent-Child Sexual Communication Questionnaire assesses youths' perceived quality and quantity of risk-specific communication with their parents.
Biological Measure of N. Gonorrhoeae Acquisition | Baseline and 6 months
  Sexually transmitted infections will be measured using biological endpoint (yes/no) to evaluate intervention effects. Participants will be screened for N. gonorrhoeae and treated if necessary at baseline. They will be tested again 12 months later to determine rate of STI acquisition.
Biological Measure of C. Trachomatis Acquisition | Baseline and 6 months
  Sexually transmitted infections will be measured using biological endpoint (yes/no) to evaluate intervention effects. Participants will be screened for C. Trachomatis and treated if necessary at baseline. They will be tested again 12 months later to determine rate of STI acquisition.
Biological Measure of T. Vaginalis Acquisition | Baseline and 6 months
  Sexually transmitted infections will be measured using biological endpoint (yes/no) to evaluate intervention effects. Participants will be screened for T. Vaginalis and treated if necessary at baseline. They will be tested again 12 months later to determine rate of STI acquisition.
Facilitator Characteristics | Baseline
  Probation teens will rate the facilitator team on similarity, credibility, competence, warmth, physical attractiveness, and sense of humor using the 9-item Perception of Peer Educator Rating Scale
Cost Effectiveness | Through study completion, an average of 2 years
  The costs associated with intervention delivery for each arm will be collected to explore differences across arms.

CONTACTS AND LOCATIONS:
Overall Officials: Geri DONENBERG, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donenberg GR, Emerson E, Mackesy-Amiti ME, Udell W. HIV-Risk Reduction with Juvenile Offenders on Probation. J Child Fam Stud. 2015 Jun 1;24(6):1672-1684. doi: 10.1007/s10826-014-9970-z. PMID 26097376
- [Background] Udell W, Donenberg G, Emerson E. Parents matter in HIV-risk among probation youth. J Fam Psychol. 2011 Oct;25(5):785-9. doi: 10.1037/a0024987. PMID 21875199
- [Background] Wilson HW, Berent E, Donenberg GR, Emerson EM, Rodriguez EM, Sandesara A. Trauma History and PTSD Symptoms in Juvenile Offenders on Probation. Vict Offender. 2013;8(4):10.1080/15564886.2013.835296. doi: 10.1080/15564886.2013.835296. PMID 24273468
- [Background] Donenberg G, Emerson E, Kendall AD. HIV-risk reduction intervention for juvenile offenders on probation: The PHAT Life group randomized controlled trial. Health Psychol. 2018 Apr;37(4):364-374. doi: 10.1037/hea0000582. Epub 2018 Feb 1. PMID 29389155
- [Background] Kendall AD, Emerson EM, Hartmann WE, Zinbarg RE, Donenberg GR. A Two-Week Psychosocial Intervention Reduces Future Aggression and Incarceration in Clinically Aggressive Juvenile Offenders. J Am Acad Child Adolesc Psychiatry. 2017 Dec;56(12):1053-1061. doi: 10.1016/j.jaac.2017.09.424. Epub 2017 Oct 5. PMID 29173739